CLINICAL TRIAL: NCT03791801
Title: Recovery From Optimal Neuromuscular Blockade in the Critically Ill: Randomized Control Trial
Brief Title: The Use of Sugammadex in the Critically Ill
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Roupen Hatzakorzian, MD, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-4576
Record Dates: First submitted 2018-12-18; First posted 2019-01-03 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Critical Illness
Keywords: sugammadex; rocuronium; critically ill
MeSH Terms: conditions — Critical Illness | interventions — Sugammadex; Neostigmine; Rocuronium; Glycopyrrolate

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neostigmine (Active Comparator): Will receive rocuronium and neostigmine (5-70microg/kg) + glycopyrrolate (10microg/kg) at train of four 1
  Interventions: Drug: Neostigmine; Drug: Rocuronium; Drug: Glycopyrrolate
- Sugammadex (Active Comparator): Will receive rocuronium and sugammadex (4mg/kg) after a successful intubation (ETT is in the trachea and secure).
  Interventions: Drug: Sugammadex; Drug: Rocuronium

INTERVENTIONS:
Drug: Sugammadex — the reversal of neuromuscular blockade with sugammadex compared to neostigmine.
  Other Names: Bridion
  Arms: Sugammadex
Drug: Neostigmine — the reversal of neuromuscular blockade with sugammadex compared to neostigmine.
  Other Names: Prostigmin
  Arms: Neostigmine
Drug: Rocuronium — Both groups will receive rocuronium for paralysis during intubation
  Other Names: Zemuron
Drug: Glycopyrrolate — The reversal of neuromuscular blockade with sugammadex compared to neostigmine/glycopyrrolate
  Other Names: Robinul
  Arms: Neostigmine

SUMMARY:
Moderate and Deep neuromuscular blockade (rocuronium administered to a train of four count 0 and post-tetanic count of 1-2) in critically ill patients needing intubation or procedures can be reversed immediately and effectively by sugammadex avoiding unnecessary paralysis in an already weakened population

DETAILED DESCRIPTION:
The Critically ill is a special population needing immediate and aggressive treatments and interventions. Neuromuscular blockade is frequently used to secure an airway, optimize ventilation/oxygenation in ARDS, aid in maintaining hypothermia in patients post-cardiac arrest. Muscle relaxants can also contribute to neuromuscular weakness in the critically ill which can be a devastating condition. Appropriate depth of neuromuscular blockade is important but unnecessary paralysis need to be avoided. Rocuronium is one of the most popular neuromuscular blockade agents used in the critically ill (1). Sugammadex is a modified γ-cyclodextrin that reverses the effect of the steroidal nondepolarizing neuromuscular blocking agents rocuronium and vecuronium (2). Sugammadex results in rapid, predictable recovery from moderate and deep neuromuscular blockade. Sugammadex has been mostly studied and used in the surgical population but its use outside the operating room is still very relevant. The investigators set up to evaluate the potential benefit that may result from the reversal of NMB with sugammadex compared to neostigmine.

Objectives

In critically ill patients undergoing intubation receiving appropriate depth of NMB (moderate and deep blockade) the investigators will assess:

Primary objective:

1. To determine if choice of reversal agent affects time from intubation to return of a train of four (TOF) count of 1, and, separately, to return of a TOF ratio >0.9

Secondary objectives:

1. To document the ability of 1.0 mg/kg rocuronium (maximum 100 mg) to achieve satisfactory intubation conditions in the ICU, based on measurement of the number of intubation attempts and intubation grades in the entire cohort
2. To document General adverse effects: Hemodynamic instability, need for vasopressors etc

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requiring intubation in the intensive care unit

Exclusion Criteria:

* Patients younger than 18 yr, to have known or suspected neuromuscular disease, allergies to medications to be used during intubation, a (family) history of malignant hyperthermia or severe renal insufficiency (glomerular filtration rate <30 ml/h) will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Train of four ratio >0.9 | up to 12 weeks
  time from intubation to return of a train of four (TOF) count of 1, and, separately, to return of a TOF ratio >0.9

CONTACTS AND LOCATIONS:
Overall Officials: Roupen Hatzakorzian, MD MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - McGill University Health Center, Montreal, Quebec
  - MUHC, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No